## Remote Neurobased Approach to Aphasia Therapy

February 24, 2022



## **Information Sheet**

- **Title of the research project**: Neurorehabilitation for Aphasia Applied in a Remote Setting
- PI: Maja From Andersen, Roc Boronat, 138 08018 Barcelona, majahaugstrupfrom.andersen01@estudiant.upf.edu
- **Institution**: Universitat Pompeu Fabra
- Objectives and duration of the project: The goal of this study is to provide a mobile application for aphasia which may facilitate recovery of language function. Therapy methods based on how the brain processes language can improve recovery for people with aphasia, and this study investigates whether therapy can be provided for the person with aphasia to practice at home with a mobile device. In order to create a therapy application, this pilot study is being done to test the usability with the application, and it will require the use of a mobile application for two weeks with completion of activities within the application every day during the two weeks.
- Methodology and participation: The application will consist of small tasks to practice language, such as naming objects and tasks involving sound, video, and images. The tasks will also require you to make voice recordings of, for example, words or short sentences. The instructions to use the application and the mobile device will be clearly explained on the first day, and afterwards you can take the device home. During the two weeks, you will be reminded two times per day to use the application. The application will collect data about when and for how long the application is used, data on the interactions, for example clicks, that you make within the application, and it will also save the voice recordings. After two weeks, you will return the mobile device and end the study. At this point, there will be a questionnaire asking about the usability of the application and the satisfaction with the process.
- **Privacy**: In order to protect your privacy, we will not identify your data with your name, but rather with a code that will only be known to the research team members. In order to make data only accessible to research team members, physical data will be stored in a locked secure location and digital data will be stored with access control systems. In the event of data publication, only anonymous data will be published. Anonymized data may be hosted or published in a public repository.
- **Risks and benefits**: Participating in this study does not entail risks greater than those ordinarily encountered in daily life. We cannot and do not guarantee that you will receive any benefits from this study.
- **Voluntary participation**: Your participation in this study is on a voluntary basis and you may withdraw from the study at any time without having to justify why.
- **Contact information**: If you have any question about this study, you may contact the PI (Maja From Andersen, <a href="majahaugstrupfrom.andersen01@estudiant.upf.edu">majahaugstrupfrom.andersen01@estudiant.upf.edu</a>),



Klaudia Grechuta (<u>kgrechuta@ibecbarcelona.eu</u>) or Javier de la Torre Costa (<u>jdelatorre@ibecbarcelona.eu</u>).

- If you have doubts, complaints, or questions about this study or about your rights as a research participant, you may contact UPF's Institutional Committee for the Ethical Review of Projects (CIREP) by phone (+34935422186) or by email (<a href="mailto:secretaria.cirep@upf.edu">secretaria.cirep@upf.edu</a>). CIREP is not part of the research team and will treat any information you send confidentially.
- In accordance with the General Data Protection Regulation (GDPR) 2016/679 (EU), we provide the following information:

**Data controller:** Universitat Pompeu Fabra. Pl. de la Mercè, 10-12. 08002 Barcelona. Tel. +34935422000. You can contact UPF's Data Protection Officer by sending an email to dpd@upf.edu.

**Purposes of the processing:** carrying out the above mentioned research project. Personal data will be kept during the execution of the project and two more years after its finalization for its scientific validation.

Legal basis: data owner's consent. You can withdraw your consent at any time.

**Recipients:** your personal data will be processed by Universitat Pompeu Fabra and Institute for Bioengineering of Catalonia (IBEC).

**Rights:** access, rectification, or erasure of your personal data, as well as data portability and the restriction or objection to the processing of your personal data. Rights may be exercised by contacting UPF's General Manager (gerencia@upf.edu). You have the right to lodge a complaint with the Catalan Data Protection Authority if you think we have not properly managed your rights.



## **Informed Consent Form**

- Title of the research project: Neurorehabilitation for Aphasia Applied in a Remote Setting
- PI: Maja From Andersen, Roc Boronat, 138 08018 Barcelona, majahaugstrupfrom.andersen01@estudiant.upf.edu
- Institution: Universitat Pompeu Fabra
- I HEREBY CONFIRM that:
  - I have read the information sheet regarding the research project,
  - I have been able to formulate any question on the project,
  - I have received enough information on the project,
  - I am between 18 and 65 years old.
- I UNDERSTAND that my participation is voluntary and that I can withdraw from or opt out of the study at any time without any need to justify my decision.

| The same of the sa |
|---|
| ☐ I GIVE MY CONSENT to participate in this study. |
| <ul> <li>I GIVE MY CONSENT to:</li> <li>i. processing of personal data in the form of voice recordings,</li> <li>ii. publication of anonymized data in an open science repository.</li> </ul> |
| Name and last name(s): |
| Signature: |
| Place and date: |

In accordance with the General Data Protection Regulation (GDPR) 2016/679 (EU), we provide the following information:

**Data controller:** Universitat Pompeu Fabra. Pl. de la Mercè, 10-12. 08002 Barcelona. Tel. +34935422000. You can contact UPF's Data Protection Officer by sending an email to dpd@upf.edu.

**Purposes of the processing:** carrying out the above mentioned research project. Personal data will be kept during the execution of the project and two more years after its finalization for its scientific validation.

Legal basis: data owner's consent. You can withdraw your consent at any time.

**Recipients:** your personal data will be processed by Universitat Pompeu Fabra and Institute for Bioengineering of Catalonia (IBEC).

**Rights:** access, rectification, or erasure of your personal data, as well as data portability and the restriction or objection to the processing of your personal data. Rights may be exercised by contacting UPF's General Manager (<a href="mailto:gerencia@upf.edu">gerencia@upf.edu</a>). You have the right to lodge a complaint with the Catalan Data Protection Authority if you think we have not properly managed your rights.